CLINICAL TRIAL: NCT01419860
Title: Evaluation of Microcirculation in Colon Wall and Bowel Anastomosis by Laser Induced Fluorescence Video Angiography of Indocyanine Green
Brief Title: Evaluation of Microcirculation in Colon Wall and Bowel Anastomosis by Laser Induced Fluorescence Video Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Microcirculation of colon
Record Dates: First submitted 2011-06-30; First posted 2011-08-18 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2015-12

CONDITIONS: Colon Cancer; Benign Colon Diseases
Keywords: Microcirculation; Colon; Anastomosis; ICG; Gastro surgery; benign colon diseases requiring resection
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pixel intensity (Experimental): Pixel intensity of fluorescence signal describing pixel microcirculation of colon
  Interventions: Procedure: Elective colon resection

INTERVENTIONS:
Procedure: Elective colon resection — In our scientific experiment, we evaluate microcirculation in colon wall and anastomosis with laser induced fluorescence videoangiography of ICG. By implementing this technique we can measure average pixel intensity of fluorescence signal in area of interest on bowel, which represents tissue perfusion in this respective part of intestinal wall.
  Other Names: Surgical colon operations; Right sided hemicolectomy; Left sided hemicolectomy; Sigmoideum resection; Subtotal colon resection

SUMMARY:
The aim of the study is to describe utility of dynamic fluorescence videoangiography of indocyanine green (ICG) in gastrointestinal surgery, for evaluation of microcirculation in colon wall and anastomosis before and after surgical resection; and if this technique can guide the surgeon to peroperative decision making considering recreate a new anastomosis or stoma for preventing anastomotic failure or stomia necrosis.

DETAILED DESCRIPTION:
In our study the investigators prospectively include patients with colon cancer requiring elective surgical operation. All types of colon resection were carried out according to standard procedures. Guidelines for preoperative examination according to NGICG (Norwegian Gastro-Intestinal Cancer Group) to grade the disease, select the most suitable patients and plan further treatment.

Microcirculation of colon wall was assessed by dynamic laser-induced-fluorescence-videoangiography (IC-VIEW, PULSION Medical Systems AG, Munich, Germany) of indocyanine green (ICG). ICG is a water-soluble tricarbocyanine dye that binds strongly to plasma proteins after intravenous injection and is exclusively distributed in intravascular space. Additionally this system houses a laser (energy Pi = 0.16 W, wavelength = 780 nm) that causes excitation/illumination of the fluorescence light from intravascular plasma bound ICG. This light has a spectral range near-infrared energy (NIR) with a maximum at 805 nm and emits fluorescence at 835 nm. It passes through infrared filter on a digital video camera and results in recording of real time fluorescent image from perfusion of plasma bound ICG within small plexus of blood vessels in the bowel wall. Besides that it also demonstrates perfusion from surrounding structures such as appendix epiploic and pericolic fat. The maximum penetration of the laser into tissue is 3-5 mm and general normal thickness of colon wall is 3-5 mm. This method makes it a presentable tracer for tissue perfusion of anterior bowel wall.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colon cancer requiring elective surgical operation.

Exclusion Criteria:

* Pregnancy
* Children or patients below the age of 18 years
* Advanced renal or hepatic failure
* Previous allergic reactions to ICG and iodide
* Chronic anemia
* Active haematologic disease
* Women of fertile age needed a negative pregnancy test to be included
* Patients with previous colectomy or anorectal surgery were also excluded due to anatomical insult on mesenterial circulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of microcirculation in colon wall and bowel anastomosis by laser induced fluorescence video angiography of indocyanine green | 2 min
  The purpose of our study is to evaluate the microcirculation in the colon wall and bowel anastomosis with laser-induced-fluorescence videoangiography of indocyanine green (ICG), before and after bowel resection.

SECONDARY OUTCOMES:
Predicting perfusion deficit with laser-induced ICG fluorescence video angiography | 2 min
  New method for predicting perfusion deficits and peroperative guide the surgeon in decision to recreate a new anastomosis or stoma.

CONTACTS AND LOCATIONS:
Overall Officials: Muiz A. Chaudhry, MD, Principal Investigator — Ostfold Hospital Trust HF
Locations (1):
- Østfold Hospital Trust HF, Fredrikstad, Østfold fylke, Norway

REFERENCES:
- [Background] Marston A. Vascular disorders of the colon. Acta Chir Belg. 1967 Dec 2;Suppl 2:80-92. No abstract available. PMID 5621502
- [Background] Massacesi AL, Sacchi L, Bergamini F, Bottoni F. The prevalence of retinal angiomatous proliferation in age-related macular degeneration with occult choroidal neovascularization. Graefes Arch Clin Exp Ophthalmol. 2008 Jan;246(1):89-92. doi: 10.1007/s00417-007-0638-x. Epub 2007 Jul 25. PMID 17653567
- [Background] Ba ZF, Yokoyama Y, Toth B, Rue LW 3rd, Bland KI, Chaudry IH. Gender differences in small intestinal endothelial function: inhibitory role of androgens. Am J Physiol Gastrointest Liver Physiol. 2004 Mar;286(3):G452-7. doi: 10.1152/ajpgi.00357.2003. Epub 2003 Oct 16. PMID 14563675
- [Background] Handa T, Katare RG, Sasaguri S, Sato T. Preliminary experience for the evaluation of the intraoperative graft patency with real color charge-coupled device camera system: an advanced device for simultaneous capturing of color and near-infrared images during coronary artery bypass graft. Interact Cardiovasc Thorac Surg. 2009 Aug;9(2):150-4. doi: 10.1510/icvts.2008.201418. Epub 2009 May 7. PMID 19423513
- [Background] Holm C, Mayr M, Hofter E, Dornseifer U, Ninkovic M. Assessment of the patency of microvascular anastomoses using microscope-integrated near-infrared angiography: a preliminary study. Microsurgery. 2009;29(7):509-14. doi: 10.1002/micr.20645. PMID 19306390
- [Background] Pena-Tapia PG, Kemmling A, Czabanka M, Vajkoczy P, Schmiedek P. Identification of the optimal cortical target point for extracranial-intracranial bypass surgery in patients with hemodynamic cerebrovascular insufficiency. J Neurosurg. 2008 Apr;108(4):655-61. doi: 10.3171/JNS/2008/108/4/0655. PMID 18377242
- [Background] Murawa D, Hirche C, Dresel S, Hunerbein M. Sentinel lymph node biopsy in breast cancer guided by indocyanine green fluorescence. Br J Surg. 2009 Nov;96(11):1289-94. doi: 10.1002/bjs.6721. PMID 19847873
- [Result] Chambers WM, Mortensen NJ. Postoperative leakage and abscess formation after colorectal surgery. Best Pract Res Clin Gastroenterol. 2004 Oct;18(5):865-80. doi: 10.1016/j.bpg.2004.06.026. PMID 15494283
- [Result] Alves A, Panis Y, Trancart D, Regimbeau JM, Pocard M, Valleur P. Factors associated with clinically significant anastomotic leakage after large bowel resection: multivariate analysis of 707 patients. World J Surg. 2002 Apr;26(4):499-502. doi: 10.1007/s00268-001-0256-4. Epub 2002 Feb 4. PMID 11910487
- [Result] Buchs NC, Gervaz P, Secic M, Bucher P, Mugnier-Konrad B, Morel P. Incidence, consequences, and risk factors for anastomotic dehiscence after colorectal surgery: a prospective monocentric study. Int J Colorectal Dis. 2008 Mar;23(3):265-70. doi: 10.1007/s00384-007-0399-3. Epub 2007 Nov 22. PMID 18034250
- [Result] Lustosa SA, Matos D, Atallah AN, Castro AA. Stapled versus handsewn methods for colorectal anastomosis surgery: a systematic review of randomized controlled trials. Sao Paulo Med J. 2002 Sep 2;120(5):132-6. doi: 10.1590/s1516-31802002000500002. PMID 12436148
- [Result] Lipska MA, Bissett IP, Parry BR, Merrie AE. Anastomotic leakage after lower gastrointestinal anastomosis: men are at a higher risk. ANZ J Surg. 2006 Jul;76(7):579-85. doi: 10.1111/j.1445-2197.2006.03780.x. PMID 16813622
- [Result] Leaper DJ. Angiography as an index of healing in experimental laparotomy wounds and colonic anastomoses. Ann R Coll Surg Engl. 1983 Jan;65(1):20-3. PMID 6186177
- [Result] Holm C, Mayr M, Hofter E, Becker A, Pfeiffer UJ, Muhlbauer W. Intraoperative evaluation of skin-flap viability using laser-induced fluorescence of indocyanine green. Br J Plast Surg. 2002 Dec;55(8):635-44. doi: 10.1054/bjps.2002.3969. PMID 12550116
- [Result] Muckle TJ. Plasma proteins binding of indocyanine green. Biochem Med. 1976 Feb;15(1):17-21. doi: 10.1016/0006-2944(76)90069-7. No abstract available. PMID 942422
- [Result] Prantl L, Schmitt S, Geis S, Tsui TY, Lamby P, Nerlich M, Kubale R, Zorger N, Herold T, Feuerbach S, Jung EM. Contrast harmonic ultrasound and indocyanine-green fluorescence video angiography for evaluation of dermal and subdermal microcirculation in free parascapular flaps. Clin Hemorheol Microcirc. 2008;38(2):105-18. PMID 18198412
- [Result] Lamby P, Prantl L, Gais S, Walter M, Bachthaler M, Nerlich M, Feuerbach S, Jung EM. Evaluation of the vascular integrity of free flaps based on microcirculation imaging techniques. Clin Hemorheol Microcirc. 2008;39(1-4):253-63. PMID 18503134
- [Result] Mitsuhashi N, Kimura F, Shimizu H, Imamaki M, Yoshidome H, Ohtsuka M, Kato A, Yoshitomi H, Nozawa S, Furukawa K, Takeuchi D, Takayashiki T, Suda K, Igarashi T, Miyazaki M. Usefulness of intraoperative fluorescence imaging to evaluate local anatomy in hepatobiliary surgery. J Hepatobiliary Pancreat Surg. 2008;15(5):508-14. doi: 10.1007/s00534-007-1307-5. Epub 2008 Oct 4. PMID 18836805
- [Result] Thoeni RF, Cello JP. CT imaging of colitis. Radiology. 2006 Sep;240(3):623-38. doi: 10.1148/radiol.2403050818. PMID 16926320
- [Result] Krasniqi A, Gashi-Luci L, Krasniqi S, Jakupi M, Hashani Sh, Limani D, Dreshaj IA. A comparison of three single layer anastomotic techniques in the colon of the rat. Int J Surg. 2009 Feb;7(1):31-5. doi: 10.1016/j.ijsu.2008.10.005. Epub 2008 Oct 18. PMID 18976973
- [Result] Ceraldi CM, Rypins EB, Monahan M, Chang B, Sarfeh IJ. Comparison of continuous single layer polypropylene anastomosis with double layer and stapled anastomoses in elective colon resections. Am Surg. 1993 Mar;59(3):168-71. PMID 8476155
- [Result] Siegel MP, Kim YL, Roy HK, Wali RK, Backman V. Assessment of blood supply in superficial tissue by polarization-gated elastic light-scattering spectroscopy. Appl Opt. 2006 Jan 10;45(2):335-42. doi: 10.1364/ao.45.000335. PMID 16422163
- [Result] Obana A, Miki T, Hayashi K, Takeda M, Kawamura A, Mutoh T, Harino S, Fukushima I, Komatsu H, Takaku Y, et al. Survey of complications of indocyanine green angiography in Japan. Am J Ophthalmol. 1994 Dec 15;118(6):749-53. doi: 10.1016/s0002-9394(14)72554-1. PMID 7977601
- See also: Literature search — http://pubmed.gov